CLINICAL TRIAL: NCT01749553
Title: Effectiveness of an 8-week Posterior Shoulder Stretch Program on Varsity-level Overhead Athletes
Brief Title: Effectiveness of an 8-week Posterior Shoulder Stretching Program on Varsity-level Overhead Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00011276; GO18000461 (Other: Faculty of Rehabilitation Medicine Internal Grant)
Record Dates: First submitted 2012-12-11; First posted 2012-12-13 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Athlete's Shoulder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- sleeper stretch (Experimental)
  Interventions: Other: Sleeper Stretch
- no intervention (No Intervention)

INTERVENTIONS:
Other: Sleeper Stretch — Posterior shoulder stretch technique
  Arms: sleeper stretch

SUMMARY:
To Determine whether an eight-week posterior shoulder stretch was effective in increasing dominant arm internal rotation(IR) and horizontal adduction (HAd) range of motion (ROM) in a group of overhead athletes identified as having tightness of their posterior shoulder structures.

ELIGIBILITY:
Inclusion Criteria:

* varsity level athletes involved in volleyball, tennis and swimming with internal rotation deficit of greater than or equal to 15 degrees

Exclusion Criteria:

* previous surgical procedure or fracture of either shoulder or presently receiving treatment for condition affecting either shoulder

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Shoulder internal rotation and horizontal adduction range of motion | 8 weeks

SECONDARY OUTCOMES:
Rate of change in internal rotation and horizontal adduction range of motion | 0 - 4 weeks and 4 - 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judy C Chepeha, PT,PhD, Principal Investigator — University of Alberta
Locations (1):
- Department of Physical Therapy, Universiy of Alberta, Edmonton, Alberta, Canada